CLINICAL TRIAL: NCT00014495
Title: Phase I/II Trial Of Sequential Therapy With Cytarabine And Bismuth-213-Labeled HuM195 (Humanized Anti-CD33) In Patients With Advanced Myeloid Malignancies
Brief Title: Chemotherapy and Monoclonal Antibody Therapy in Treating Patients With Advanced Myeloid Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00-117; MSKCC-00117; NCI-H01-0071
Record Dates: First submitted 2001-04-10; First posted 2003-01-27 (Estimated); Results first posted 2016-01-22 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2015-12

CONDITIONS: Leukemia; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms
Keywords: recurrent childhood acute myeloid leukemia; recurrent adult acute myeloid leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; untreated adult acute myeloid leukemia; untreated childhood acute myeloid leukemia and other myeloid malignancies; refractory anemia with excess blasts; refractory anemia with excess blasts in transformation; chronic myelomonocytic leukemia; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; childhood chronic myelogenous leukemia; atypical chronic myeloid leukemia, BCR-ABL1 negative; myelodysplastic/myeloproliferative neoplasm, unclassifiable; adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with t(15;17)(q22;q12); childhood myelodysplastic syndromes
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Leukemia, Myeloid, Acute; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Anemia, Refractory, with Excess of Blasts; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Myeloproliferative Disorders; Congenital Abnormalities | interventions — Filgrastim; Cytarabine

ARMS (1):
- bismuth Bi 213 monoclonal antibody M195 & cytarabine (Experimental): Patients receive cytarabine IV continuously on days 1-5. Beginning between days 7 and 14, patients receive Bi213 MOAB M195 IV over 5 minutes up to 4 times daily over 1-4 days. Patient also receive filgrastim (G-CSF) subcutaneously daily beginning 24 hours after the final Bi213 MOAB M195 infusion and continuing until blood counts recover. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3 to 6 patients receive escalating doses of Bi213 MOAB M195 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, subsequent patients are treated at the MTD.
  Patients are followed twice weekly for 4 weeks and then monthly for 3 months
  Interventions: Biological: filgrastim; Drug: cytarabine; Radiation: bismuth Bi213 monoclonal antibody M195

INTERVENTIONS:
Biological: filgrastim
Drug: cytarabine
Radiation: bismuth Bi213 monoclonal antibody M195

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining monoclonal antibody therapy with chemotherapy may kill more cancer cells.

PURPOSE: Phase I/II trial to study the effectiveness of combining chemotherapy and monoclonal antibody therapy in treating patients who have advanced myeloid cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of bismuth Bi 213 monoclonal antibody M195 following cytarabine in patients with advanced myeloid malignancies.
* Determine the antileukemic effects of this treatment in this patient population.
* Determine the toxicity of this treatment in this patient population.
* Determine the complete remission rate of patients treated with this treatment regimen.

OUTLINE: This is a dose escalation study of bismuth Bi 213 monoclonal antibody M195 (Bi213 MOAB M195).

Patients receive cytarabine IV continuously on days 1-5. Beginning between days 7 and 14, patients receive Bi213 MOAB M195 IV over 5 minutes up to 4 times daily over 1-4 days. Patient also receive filgrastim (G-CSF) subcutaneously daily beginning 24 hours after the final Bi213 MOAB M195 infusion and continuing until blood counts recover. Treatment continues in the absence of disease progression or unacceptable toxicity.

Cohorts of 3 to 6 patients receive escalating doses of Bi213 MOAB M195 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, subsequent patients are treated at the MTD.

Patients are followed twice weekly for 4 weeks and then monthly for 3 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* One of the following diagnoses:

  * Pathologically confirmed acute myeloid leukemia (AML) meeting one of the following criteria:

    * Newly diagnosed AML, over age 60, and not eligible for higher priority protocols
    * Newly diagnosed AML and unable to receive anthracycline-containing or high-dose cytarabine-containing regimens
    * AML in relapse
    * AML refractory to two courses of standard induction chemotherapy or one course of high-dose cytarabine-containing induction chemotherapy
  * Chronic myelogenous leukemia in accelerated phase or myeloid blast crisis
  * Refractory anemia with excess blasts (RAEB), RAEB in transformation, or chronic myelomonocytic leukemia
* More than 25% of bone marrow blasts must be CD33 positive
* Not a candidate for immediate bone marrow transplantation with a HLA-compatible donor
* No active CNS leukemia

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* Karnofsky 60-100%

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin no greater than 2 mg/dL (unless due to leukemia or Gilbert's disease)
* Alkaline phosphatase no greater than 2.5 times upper limit of normal (ULN)
* AST no greater than 2.5 times ULN

Renal:

* Creatinine less than 2 mg/dL OR
* Creatinine clearance greater than 60 mL/min

Cardiovascular:

* No New York Heart Association class III or IV cardiac disease

Pulmonary:

* No pulmonary disease

Other:

* No detectable antibodies to monoclonal antibody M195
* No serious active uncontrolled infection
* No other concurrent active malignancy requiring therapy
* No other serious or life-threatening conditions that would preclude study
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 3 weeks since prior biologic therapy and recovered

Chemotherapy:

* See Disease Characteristics
* Prior hydroxyurea allowed if discontinued before study treatment
* At least 3 weeks since other prior chemotherapy and recovered

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 3 weeks since prior radiotherapy and recovered

Surgery:

* Not specified

Max Age: 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2000-11; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph G. Jurcic, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan - Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Result] Rosenblat TL, McDevitt MR, Mulford DA, Pandit-Taskar N, Divgi CR, Panageas KS, Heaney ML, Chanel S, Morgenstern A, Sgouros G, Larson SM, Scheinberg DA, Jurcic JG. Sequential cytarabine and alpha-particle immunotherapy with bismuth-213-lintuzumab (HuM195) for acute myeloid leukemia. Clin Cancer Res. 2010 Nov 1;16(21):5303-11. doi: 10.1158/1078-0432.CCR-10-0382. Epub 2010 Sep 21. PMID 20858843
- [Result] Mulford DA, Pandit-Taskar N, McDevitt MR, et al.: Sequential therapy with cytarabine and bismuth-213 (213Bi)-labeled-HuM195 (Anti-CD33) for acute myeloid leukemia (AML). [Abstract] Blood 104 (11): A-1790, 2004.

RESULTS

PARTICIPANT FLOW:
Groups:
- Bismuth-labeled HuM195 (0.5 mCi/kg); Bismuth-labeled HuM195 (0.75 mCi/kg); Bismuth-labeled HuM195 (1 mCi/kg); Bismuth-labeled HuM195 (1.25 mCi/kg): Patients receive cytarabine IV continuously on days 1-5. Beginning between days 7 and 14, patients receive Bi213 MOAB M195 IV over 5 minutes up to 4 times daily over 1-4 days. Patient also receive filgrastim (G-CSF) subcutaneously daily beginning 24 hours after the final Bi213 MOAB M195 infusion and continuing until blood counts recover. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3 to 6 patients receive escalating doses of Bi213 MOAB M195 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, subsequent patients are treated at the MTD.
Period: Overall Study
Arm/Group | Bismuth-labeled HuM195 (0.5 mCi/kg) | Bismuth-labeled HuM195 (0.75 mCi/kg) | Bismuth-labeled HuM195 (1 mCi/kg) | Bismuth-labeled HuM195 (1.25 mCi/kg)
Started | 3 | 3 | 20 | 6
Completed | 3 | 3 | 19 | 5
Not Completed | 0 | 0 | 1 | 1
Not completed — Death | 0 | 0 | 1 | 0
Not completed — Clinical deterioration | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bismuth-labeled HuM195 (0.5 mCi/kg) | Bismuth-labeled HuM195 (0.75 mCi/kg) | Bismuth-labeled HuM195 (1 mCi/kg) | Bismuth-labeled HuM195 (1.25 mCi/kg) | Total
Number analyzed (Participants) | 3 | 3 | 20 | 6 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 9 | 1 | 14
  >=65 years | 1 | 1 | 11 | 5 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 8 | 1 | 10
  Male | 3 | 2 | 12 | 5 | 22
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 20 | 6 | 32

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose
Description: The maximum tolerated dose of bismuth Bi 213 monoclonal antibody M195 following cytarabine in patients with advanced myeloid malignancies.
Time Frame: 2 years
Measure: Number; unit: mCi/kg
Groups:
- Bismuth Bi 213 Monoclonal Antibody M195 & Cytarabine: Patients receive cytarabine IV continuously on days 1-5. Beginning between days 7 and 14, patients receive Bi213 MOAB M195 IV over 5 minutes up to 4 times daily over 1-4 days. Patient also receive filgrastim (G-CSF) subcutaneously daily beginning 24 hours after the final Bi213 MOAB M195 infusion and continuing until blood counts recover. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3 to 6 patients receive escalating doses of Bi213 MOAB M195 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, subsequent patients are treated at the MTD.
  Patients are followed twice weekly for 4 weeks and then monthly for 3 months
  filgrastim
  cytarabine
  bismuth Bi213 monoclonal antibody M195
Arm/Group | Bismuth Bi 213 Monoclonal Antibody M195 & Cytarabine
Number analyzed (Participants) | 20
mCi/kg | 1

ADVERSE EVENTS:
Arm/Group | Bismuth-labeled HuM195 (0.5 mCi/kg) | Bismuth-labeled HuM195 (0.75 mCi/kg) | Bismuth-labeled HuM195 (1 mCi/kg) | Bismuth-labeled HuM195 (1.25 mCi/kg)
Serious Adverse Events (participants affected / at risk) | 2/3 | 2/3 | 3/20 | 3/6
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 17/20 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bismuth-labeled HuM195 (0.5 mCi/kg) (N=3) | Bismuth-labeled HuM195 (0.75 mCi/kg) (N=3) | Bismuth-labeled HuM195 (1 mCi/kg) (N=20) | Bismuth-labeled HuM195 (1.25 mCi/kg) (N=6)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bismuth-labeled HuM195 (0.5 mCi/kg) (N=3) | Bismuth-labeled HuM195 (0.75 mCi/kg) (N=3) | Bismuth-labeled HuM195 (1 mCi/kg) (N=20) | Bismuth-labeled HuM195 (1.25 mCi/kg) (N=6)
Creatinine increased (Investigations) | 1 (2) | 0 (0) | 4 (7) | 1 (1)
Derm, skin other (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (3) | 1 (1) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 1 (2) | 10 (58) | 2 (5)
Infection, other (Infections and infestations) | 1 (1) | 3 (5) | 14 (28) | 3 (6)
White blood cell decreased (Investigations) | 2 (8) | 3 (6) | 15 (106) | 6 (46)
Neutrophil count decreased (Investigations) | 1 (2) | 2 (9) | 7 (18) | 4 (13)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (4)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 2 (15) | 12 (83) | 4 (36)
Alkaline phosphatase increase (Investigations) | 0 (0) | 0 (0) | 4 (6) | 0 (0)
Allergic Reaction (Immune system disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Blood bilirubin increase (Investigations) | 0 (0) | 0 (0) | 7 (34) | 3 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Fever (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Hemorrhage, other (General disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 3 (3)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (4)
Rigors, chills (General disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Aspartate aminotransferase increase (Investigations) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Alanine aminotransferase increase (Investigations) | 0 (0) | 0 (0) | 6 (13) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Adult Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes